CLINICAL TRIAL: NCT03051919
Title: Staple Line Reinforcement Methods in Laparoscopic Sleeve Gastrectomy: Comparison of Burst Pressures and Leaks
Brief Title: Reinforcement Method in Laparoscopic Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, M.Timucin Aydin, Attending Surgeon, Department of Surgery, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMTRH
Record Dates: First submitted 2015-04-01; First posted 2017-02-14 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Laparoscopic Sleeve Gastrectomy
Keywords: Laparoscopic sleeve gastrectomy; reinforcement; leak
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — resected stomachs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- no reinforcement: Group I: 25 patients; no reinforcement (NoR) Observation : Patients would be followed up for any signs of leaks. If any, treatment would be offered appropriataly but the results of treatment are not affiliated as a part in the study.
  Interventions: Other: observation
- fibrin glue: Group II: 26 patients; fibrin glue (FG) Observation : Patients would be followed up for any signs of leaks. If any, treatment would be offered appropriataly but the results of treatment are not affiliated as a part in the study.
  Interventions: Other: observation
- suture reinforcement: Group III: 44 patients; suture reinforcement with 2-0 polypropylene suture (S) Observation : Patients would be followed up for any signs of leaks. If any, treatment would be offered appropriataly but the results of treatment are not affiliated as a part in the study.
  Interventions: Other: observation
- biological buttressing materaia: Group IV: 14 patients; biological buttressing material Observation : Patients would be followed up for any signs of leaks. If any, treatment would be offered appropriataly but the results of treatment are not affiliated as a part in the study.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation

SUMMARY:
Laparoscopic sleeve gastrectomy is a technically simple popular bariatric operation with acceptable results. Leaks can occur in long staple lines; therefore, variable reinforcement methods are used.

DETAILED DESCRIPTION:
The investigator compared non-reinforced stapling with three staple line reinforcement methods (suturing, absorbable buttressing material and fibrin glue) in laparoscopic sleeve gastrectomy.

The resected stomach specimens were treated in the same manner of reinforcement as used in the surgeries of the corresponding patients and then insufflated until a burst occurred. The burst pressures of the resected stomach specimens and postoperative events of the patients were recorded.

ELIGIBILITY:
Inclusion Criteria:

* body mass index >40 kg/m2

Exclusion Criteria:

* disruption of the resected stomach during extraction from the abdomen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 118 patients with body mass index >40 kg/m2 underwent sleeve gastrectomy and were enrolled into four groups
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
assessing prevalence of leaks among different reinforcement methods | 3 months
  observation

IPD SHARING:
Plan to Share IPD: Undecided